CLINICAL TRIAL: NCT05828355
Title: Effectiveness of the KC@H Programme Compared With Clinic-based Rehabilitation in Patients Recovering From Anterior Cruciate Ligament Reconstruction: Study Protocol for a Single-centre, Randomised Controlled Superiority Trial.
Brief Title: The Knee Care @Home Programme Following Anterior Ligament Reconstruction
Acronym: KC@H
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Évora (Other)
Collaborators: Comprehensive Health Research Center (Other); Fundação para a Ciência e a Tecnologia (Other); Hospital da Misericórdia de Évora (Unknown)
Responsible Party: Principal Investigator, Joao Paulo Brites de Sousa, Assistant Professor, University of Évora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KC@H RCT
Record Dates: First submitted 2023-03-17; First posted 2023-04-25 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Anterior Cruciate Ligament Reconstruction; Patient-reported Outcomes Measures; Clinician-reported Outcomes Measures; Functional Performance; Clinical Relevance; Internet-based Intervention; Exercise Therapy
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinic-based Rehabilitation (No Intervention): Individualised clinic-based face-to-face sessions with a physiotherapist in public or private rehabilitation facility
- Knee Care@Home (Experimental): Individualised synchronous internet-based remote sessions at home via conferencing software under the supervision of a certified exercise and health coach as a complement to conventional clinic-based rehabilitation sessions.
  Interventions: Other: Knee Care@Home Programme

INTERVENTIONS:
Other: Knee Care@Home Programme — Over 24 weeks after undergoing surgical reconstruction of the anterior cruciate ligament, patients in the intervention group will receive supervised guidance on therapeutic exercises to be performed at home. This guidance will be provided through individualised synchronous internet-based remote sessions using conferencing software.
  Other Names: Synchronous internet-based remote sessions; Therapeutic Exercise
  Arms: Knee Care@Home

SUMMARY:
Background: Patients who are unable to fully comply with conventional clinic-based rehabilitation sessions after anterior cruciate ligament reconstruction may find additional internet-based sessions beneficial. These remote sessions include therapeutic exercises that can be done at home, potentially extending the reach of rehabilitation services to underserved areas, prolonging the duration of care, and providing improved supervision.

Objective: To determine if the Knee Care at Home programme is more effective than conventional clinic-based rehabilitation alone in improving patient-reported, clinician-reported, and physical functional performance outcome measures after anterior cruciate ligament reconstruction. Additionally, the trial pursues to assess the significance of changes in outcome measures for clinical practice.

Methods/design: This protocol outlines a randomised controlled trial for postoperative recovery following anterior cruciate ligament reconstruction. Adult participants of both sexes who meet specific criteria will be randomly assigned to either the Clinic-based Rehabilitation group or the Knee Care at Home group. Only the latter group will receive internet-based sessions of therapeutic exercises at home, in addition to clinic-based rehabilitation sessions. A follow-up evaluation will be conducted for both groups 12 weeks after the intervention ends.

Expected Results: The Knee Care at Home programme is superior to conventional clinic-based rehabilitation alone for patients recovering from anterior cruciate ligament reconstruction across multiple outcome measures. Also, the programme has the potential to promote superior recovery and extend the reach and duration of care.

ELIGIBILITY:
Inclusion Criteria:

* Undergone primary ACLR regardless of surgical method and choice of autograft.
* Have a healthy contralateral (opposite) knee.
* The time between ACL injury and ACLR should not exceed 12 months.

Exclusion Criteria:

* Declined to participate.
* Concomitant osteochondral injuries.
* Undergone multiple reconstructions of the lateral collateral ligament or posterior cruciate ligament.
* Significant lower limb injuries within the 12 months before the ACL injury.
* Medical conditions that may affect recovery.
* Using medication for mental health disorders.
* Severe impairments in communication or balance.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Standing height | Preoperative consultation
  Patients are measured for standing height in centimetres using a stadiometer placed against the wall. They are instructed to stand with their backs against the wall, heels together, head in a natural position, legs straight, arms at their sides, and shoulders relaxed. They should not wear shoes or heavy clothing that could affect their height measurement. The measurement arm is lowered to rest gently on the patient's head, and the measurement is rounded off to the nearest decimal.
Weight | up to 36 weeks postoperative
  Patients are assessed for weight (body mass in kilograms) using a traditional weighing scale. The scale is placed on a flat and stable surface, and patients are advised not to wear shoes or heavy clothing that could affect their weight measurement. They are instructed to stand still in the centre of the scale, with their feet evenly positioned and their weight evenly distributed. The weight measurement is then recorded and rounded off to the nearest decimal.
Knee pain during the last 24 hours | up to 36 weeks postoperative
  Visual Analogue Scale (VAS). Patients provide feedback on the intensity of their knee pain by marking a point on a 100mm straight horizontal line. The beginning of the line represents "no pain" while the end represents the "worst possible pain". A ruler is used to measure the distance (in millimetres) from 0 to the patient's marking. Additionally, a numerical value and Wong-Baker faces scale will be presented to the patient for reference.
Knee pain during the last week | up to 36 weeks postoperative
  Knee Injury and Osteoarthritis Outcome Score (KOOS) for pain. Patients provide feedback on the severity of their knee pain using a standard 5-point Likert scale. Each response option is assigned a numerical value (0 for none, 1 for mild, 2 for moderate, 3 for severe, and 4 for extreme). A score of 0 indicates no pain, while a score of 32 (based on 8 questions) indicates extreme pain.
Knee symptoms and stiffness during the last week | up to 36 weeks postoperative
  Knee injury and Osteoarthritis Outcome Score (KOOS) for symptoms and stiffness. Patients are asked to rate their knee symptoms and stiffness using a standard 5-point Likert scale, with each response option assigned a numerical value (0, 1, 2, 3, 4). A score of 0 indicates total absence of symptoms, while a score of 20 (based on 5 questions) indicates constant symptoms. For knee stiffness, a score of 0 indicates total absence, while a score of 8 (based on 2 questions) indicates extreme stiffness.
Knee-related physical function during the last week | up to 36 weeks postoperative
  Knee Injury and Osteoarthritis Outcome Score - Physical Function Short Form (KOOS-PS). Patients use a standard 5-point Likert scale to provide feedback on their knee-related physical function. Each response option is assigned a numerical value (0 for none, 1 for mild, 2 for moderate, 3 for severe, and 4 for extreme). A score of 0 indicates no difficulties, while a score of 28 (based on 7 questions) indicates extreme difficulties.
Knee function in daily living, sports, and recreational activities during the last week | up to 36 weeks postoperative
  Knee injury and Osteoarthritis Outcome Score (KOOS) for function in daily living, sports, and recreational activities: Patients are asked to rate their knee function in daily living, sports, and recreational activities using a standard 5-point Likert scale. Each response option is given a numerical value (0 for none, 1 for mild, 2 for moderate, 3 for severe, and 4 for extreme). For knee function in daily living, a score of 0 indicates no difficulties, while a score of 68 (based on 17 questions) indicates extreme difficulties. Similarly, for knee function in sports and recreational activities, a score of 0 indicates no difficulties, while a score of 20 (based on 5 questions) indicates extreme difficulties.
Knee-related quality of life | up to 36 weeks postoperative
  Knee injury and Osteoarthritis Outcome Score (KOOS) for quality of life. Patients using a standard 5-point Likert scale to provide feedback on their knee-related quality of life. Each response option is given a numerical value (0, 1, 2, 3, 4) and a raw score is determined based on their responses. A score of 0 indicates no impact, while a score of 4 (based on 4 questions) indicates extreme impact on the quality of life.
Knee joint effusion | up to 36 weeks postoperative
  Patellar Tap/Ballottement Test. Patients are evaluated for knee effusion while lying supine on an examination table. The assessor applies downward strokes from the thigh to the leg with the non-dominant hand and then grasps the upper portion of the knee just above the patella. Using two fingers of the dominant hand they press the patella against the femur in a posterior direction. A positive test result for knee effusion is indicated by increased patellar waving or a spongy joint sensation. The test is then repeated on the opposite knee for comparison.
Passive knee flexion and extension range of motion | up to 36 weeks postoperative
  Hand-held Goniometry (HHG): Passive knee extension and flexion range of motion are measured using a long-arm goniometer. The goniometer axis is placed at the lateral epicondyle of the femur. The proximal arm is placed alongside the lateral midline of the femur, using the greater trochanter as a reference, while the distal arm is placed alongside the lateral midline of the fibula, using the lateral malleolus and fibular head as references. Passive knee flexion: the patient lies in a supine position on the table with the lower limbs in an anatomical position. The assessor flexes the knee by sliding the patient's foot along the table towards the pelvis and then taking the passive range of motion measurement. Passive knee extension: the patient lies in a supine position on the table with a towel under the ankle with the knee extended as far as possible. The assessor provides added pressure to the knee in the direction of extension and then takes the passive range of motion measurement.
Knee extensor and flexor muscle length | up to 36 weeks postoperative
  Hand-held Goniometry (HHG): The length of the knee flexors and extensors muscles is measured with a long-arm goniometer. The goniometer axis placed at the lateral epicondyle of the femur. For the flexor muscle length, the patient lies in a prone position with both hips of the lower extremity extended on the table, and the knee to be tested moves to maximal achieved flexion, and the measurement of knee flexion is taken (test side). For the extensors length, the patient lies in a supine position with the hip of the lower extremity to be measured in 90 degrees of flexion on the table. While the assessor helps to maintain the hip position, the patient executes a knee extension, and the measurement of knee flexion is taken (test side).
Knee extensor and flexor isometric muscle strength | up to 36 weeks postoperative
  Hand-held Dynamometry (HHD): The microFET®2 is used to measure the isometric strength of the hamstrings and quadriceps in patients. This measurement is taken on both knees to allow for comparison. The patient is seated with their hips and knees flexed at a 90-degree angle on an examination table. The assessor stabilizes the patient's leg using the leg of the examination table as support for the hand-held dynamometer. The patient is then instructed to apply maximum force against the device. First, the patient is asked to try to extend the knee, and then they are asked to flex the knee. Three repetitions are performed for both extension and flexion.
Knee pain catatrophising | up to 36 weeks postoperative
  Pain Catastrophizing Scale (PCS): Patients are asked to provide feedback on their thoughts, feelings, or perceptions related to pain using a standard 5-point Likert scale. Each response option is assigned a numerical value (0 for "not at all", 1 for "a slight degree", 2 for "moderate degree", 3 for "great degree", to 4 for "all the time"). A score of 0 indicates a total absence of catastrophic thinking, while a score of 52 (based on 13 questions) indicates a persistent tendency towards catastrophising thoughts about pain.
Anxiety, depression, and stress during last week | up to 36 weeks postoperative
  Depression Anxiety Stress Scales (DASS-21) short-form: Patients use a standard 4-point Likert scale. Each response option is assigned a numerical value (0 for "did not apply to me at all", 1 for "applied to me to some degree, or some of the time", 2 for "applied to me to a considerable degree or a good part of time", and 3 for "applied to me very much or most of the time"). Cut-off scores determine the severity. For depression, based on 7 items, scores of 0 to 9 are considered normal, 10 to 13 are mild, 14 to 20 are moderate, 21 to 27 are severe, and 28 or higher are extremely severe. For anxiety, based on 7 items, scores of 0 to 7 are normal, 8 to 9 are mild, 10 to 14 are moderate, 15 to 19 are severe, and 20 or higher are extremely severe. For stress, based on 7 items, scores of 0 to 14 are normal, 15 to 18 are mild, 19 to 25 are moderate, 26 to 33 are severe, and 34 or higher are extremely severe.
Hop distance on a single leg | up to 36 weeks postoperative
  Patients are instructed to stand on the leg being tested, hop, and then land on the same limb, jumping as far as possible. The distance hopped is measured at the level of the great toe and recorded to the nearest centimetre using a standard measuring tape that is fixed to the floor. Both lower limbs are evaluated for comparison.
Ability to ascend and descend a flight of stairs (12 steps) | up to 36 weeks postoperative
  Stair Climbing (SC) test: Patients will be timed as they ascend and descend a flight of 12 stairs as quickly as possible. The number of steps they perform in 30-second intervals will also be counted.

SECONDARY OUTCOMES:
Symptom State | up to 36 weeks postoperative
  Patient Acceptable Symptomatic State (PASS): Patients provide their perspectives on the final PROM scores, which indicate their satisfaction with symptoms. For each PROM score, patients are asked a question with the answer option "yes" or "no".
Clinical Benefit | up to 36 weeks postoperative
  Substantial Clinical Benefit (SCB): Patients are surveyed to gather their perspective on the change in PROM scores that indicates a significant or optimal improvement. For each change in score, patients are asked a question with answer options displayed on a 7-point Likert scale, ranging from "significant and marked improvement" to "no improvement at all".
Clinical Difference | up to 36 weeks postoperative
  Minimal Clinically Important Difference (MCID): The patients will be asked about their opinion on the minimum change in PROM scores that would show a meaningful improvement in their condition. We will use an anchor-based technique to determine the MCID.

CONTACTS AND LOCATIONS:
Overall Officials: João Paulo Sousa, PhD, Principal Investigator — Universidade de Évora - Comprehensive Health Research Center
Locations (1):
- Hospital da Misericórdia de Évora, Evora, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alegrete J, Batalha N, Fernandes O, Parraca JA, Rodrigues AM, Londral AR, Sousa JP. Effectiveness of the KC@H programme compared with clinic-based rehabilitation in patients recovering from ACL reconstruction: a study protocol for a single-centre, two-arm, single-blinded, randomised controlled superiority trial. BMJ Open Sport Exerc Med. 2024 Feb 21;10(1):e001868. doi: 10.1136/bmjsem-2023-001868. eCollection 2024. PMID 38390383